## Parental stress and disability. A psychological flexibility training programme

ID: CIPI/21/091

Document date: 15th November 2021

IP: Francisco Montesinos, Ph.D.

Study Protocol and Statistical Analysis Plan

## **Study Protocol:**

- Objective: To study the efficacy of a group treatment based on Acceptance and Commitment Therapy on parental stress in relatives of people with intellectual disabilities.
- Design: Randomized clinical trial
- Methods.

After being informed about the study, all patients giving written informed consent will be assessed to determine eligibility for study entry. Parents who meet eligibility requirements will be assessed through a standardized questionnaires, self-report instruments and randomized assigned to a waiting list or treatment.



Participants assigned to treatment arm will receive psychological intervention consistent in a 3-session group ACT-based treatment in the in a room of the collaborating NGO by a psychologist trained in third-generation therapies and experienced in working with families

Standardized questionnaires were administered before the intervention (pre-treatment), one week after its completion (post-treatment), and three months later (follow-up). Participants completed daily self-monitoring from one week before the intervention (forming the BL) until one week after the intervention, obtaining 4 measures. In addition, participants filled in their workbooks in each session

## **Intervention protocol.**

Session 1. Introducing ACT therapy. Promoting creative hopelessness: an experiential exercise to assess the effectiveness of stress coping repertoires through "Man in the hole" metaphor (Hayes et al., 2014). Training in self as context through the "Observer exercise" (Hayes et al., 2014). Homework: implementing committed actions and self-report.

Session 2. Training in values and commitment action through experiential exercises: 1) What kind of mother or father do I want to be? 2) What can I do this week to move towards the kind of parent I want to be? 3) Clarifying values about family/parenting; assessing the importance and value orientation on a scale of 0 to 10. Training in self as context through the "Observer exercise" (Hayes et al., 2014). Training in acceptance, defusion and contact with the present moment through experiential exercises: 1) Emotion Mindfulness through physicalization (Harris, 2019) 2) "Joe the Bum" metaphor (Hayes et al., 2014) and 3) "Passengers on the Bus" metaphor (Hayes et al., 2014). Homework: implementing committed actions and self-report. Homework: What can I do this week to move towards the kind of parent I want to be? Practicing Mindful breathing exercise (audio recording) and self-report.

Session 3. Training in values and commitment action through experiential exercises: 1) Identifying valuable actions in the presence of internal and external barriers. 2) Experiential exercise: "When...Then". 3) "The choice point" (Harris, 2019) 4) Our values as parents. Sharing the values on which I articulate my actions. Training in self as context through the "Observer exercise" (Hayes et al., 2014). Training in acceptance, defusion and contact with the present moment through experiential exercises: 1) Mindful breathing exercise (audio re-cording) 2) "Passengers on the Bus" metaphor (Hayes et al., 2014). Homework: implementing committed actions and self-report. Provision of support and supplementary materials.

## Statistical Analysis Plan (SAP):

The results will be analysed through non-parametric techniques (comparisons of pre, post and follow-up group means). An analysis of variance will be performed to determine the specific weight of each independent variable, as well as the possible interaction between them. The statistical approach of Jacobson and Truax (1991) will be used to estimate the clinical significance of the effect. Finally, the change in self-monitoring will be analysed through repeated measures ANOVA.